CLINICAL TRIAL: NCT00290953
Title: A Double Blind, Randomized, Phase II-III Maintenance Study of SR48692 Versus Placebo in Patients With Extensive Stage Small Cell Lung Cancer Following a First Line Chemotherapy With Cisplatin + Etoposide
Brief Title: Evaluation of the Overall Survival of Meclinertant Versus Placebo After a First Line Chemotherapy With Cisplatin + Etoposide
Acronym: SESAME
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC3679
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Lung Cancer; Pulmonary Neoplasms; Small Cell Lung Cancer
Keywords: Metastases
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma; Neoplasm Metastasis | interventions — SR 48692

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SR48692

SUMMARY:
To demonstrate an increase in overall survival for patients with newly diagnosed extended stage small cell lung cancer when treated with SR48692 versus placebo, after an initial response (complete or partial response or stable) to first line cisplatin plus etoposide.

Primary objective: comparison of overall survival between patients in the control arm and the meclinertant arm.

Secondary objectives: comparison of the progression free survival, the time to progression, the clinical benefit, the quality of life, the toxicity and safety between patients in the control arm and the meclinertant arm.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis: Histologically or cytologically proven SCLC.
* Disease stage: extensive stage
* Measurable disease by the RECIST criteria is required. Lesions that are present in previously irradiated area are non-measurable unless they have appeared or progressed since completion of the radiation.
* Radiotherapy, if applicable, must have been completed at least 4 weeks before treatment under this protocol and the subject must have recovered from any acute toxicities of radiation.
* Recovered from any surgical procedure(s).
* Calculated creatinine clearance > 55 ml/min using the Cockcroft-Gault formula: Cr Cl in ml/min = (140-age) X (weight in kg) X (1.0 for men or 0.85 for women) / (72 X serum Cr in mg/dl).
* Total bilirubin < two times the upper limit of the normal range at the institution and SGOT/AST < two times the upper limit of normal unless liver metastases are present.
* ANC > 1.5 x 109/L and platelet count > 100 x 109/L.
* Age >18 years.
* Karnofsky Performance Status > 70% .
* Subjects with no prior malignancy, or subjects with cured malignancies other than SCLC if: a) they are alive without disease recurrence for at least 5 years from the date of pathological diagnosis, and b) clinical expectation of disease recurrence is < 5% as documented in the medical record by the responsible physician, and c) they have not received any platinum-based therapy. Subjects with basal cell carcinoma or carcinoma in situ of the cervix may be eligible if adequately treated and clinical expectation of disease recurrence is < 5% as documented in the medical record by the responsible physician.
* Infertile subjects or fertile subjects who use a medically acceptable contraceptive throughout the treatment period and for 3 months following cessation of treatment. Women of childbearing potential must have documentation of a negative, serum HCG pregnancy test. Subjects must be made aware, before entering this trial, of the risk in becoming pregnant or in fathering children.
* Signed written informed consent (approved by the Ethics Committee) obtained prior to study entry.

Exclusion Criteria:

* Limited disease.
* Symptomatic brain metastases: a patient with brain and/or leptomeningeal metastases on computer tomography (CT) or Magnetic Resonance Imaging (MRI) scan may be included only if he/she is asymptomatic on neurologic exam and is not receiving corticosteroid therapy to control symptoms.
* Concurrent active cancer, including cancer stable on adjuvant therapy.
* Prior immunotherapy, biological therapy or chemotherapy for SCLC.
* Radiotherapy: Prior radiation to non-symptomatic or non-life-threatening sites.Prior radiation therapy to all potential indicator lesions. Prior radiation therapy to some but not all indicator lesions is allowed.
* Class III or IV congestive heart failure according to the New York Heart Association Classification.
* History of allergic reactions to appropriate diuretics or antiemetics (e.g., 5-HT3 antagonists) to be administered in conjunction with protocol-directed chemotherapy.
* Uncontrolled intercurrent illness.
* Lactating or pregnant women.
* Received any investigational drug within 30 days before beginning treatment with study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2002-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
- Overall survival (OS)

SECONDARY OUTCOMES:
- Progression Free Survival (PFS)
- Time to Progression (TTP)
- Clinical Benefit assessed by Performance Status and body weight
- Quality of Life using the LCSS and EuroQoL validated instruments
- Toxicity and safety assessment using NCI CTC version 2.0

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (14):
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-aventis adminsitrative office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com